CLINICAL TRIAL: NCT01474850
Title: Thoraco-abdominal Volume Variation During Recovery From Total Intravenous Anesthesia Studied by Opto-electronic Plethysmography (OEP).
Brief Title: Thoraco-abdominal Volume Variations During Anesthesia Studied by OEP.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Peter Kostic, Staff anesthesiologist, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Uppsala 2011 - 190
Record Dates: First submitted 2011-11-08; First posted 2011-11-18 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Mechanical Ventilation
Keywords: mechanical ventilation; pressure control ventilation; lung recruitment; positive end expiratory pressure; opto-electronic plethysmography; chest wall volume variation; intravenous anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- open lung (Active Comparator): The lung recruitment maneuver (RM) immediately after intubation using pressure controlled ventilation, increase in peak inspiratory pressure up to 30 cm H2O during tidal ventilation, respiratory rate 4/min and positive end expiratory pressure (PEEP) 15 cm H20. PEEP 7 cm H2O until extubation. Inspiratory oxygen concentration (FiO2) 40% during recovery from anesthesia.
  Interventions: Procedure: lung recruitment maneuver
- control (No Intervention): No recruitment maneuver is performed. PEEP 0 cm H2O. Inspiratory oxygen concentration (FiO2) 100 % during recovery from anesthesia.

INTERVENTIONS:
Procedure: lung recruitment maneuver — RM: peak inspiratory pressure 30 cmH2O, PEEP 15 cm H20 FiO2 0,4 (from end of surgery till extubation)
  Arms: open lung

SUMMARY:
The aim of this study is to examine chest wall volume changes monitored by opto-electronic plethysmography during recovery from anesthesia and early postoperative period.

DETAILED DESCRIPTION:
This is prospective, randomized clinical trial in subjects undergoing elective surgery requiring general anesthesia.

Opto-electronic plethysmography (OEP) has been developed as a non-invasive method for the analysis of chest wall motion, allowing highly accurate measurements of chest wall volume changes of different respiratory compartments in various conditions.

The investigators set out to use this technology to study chest wall volume changes during recovery from total intravenous anesthesia (from discontinuing the anesthetic agent till extubation) and early postoperative period.

The study protocol compares two different approaches:

1. The group receiving recruitment maneuver (RM) immediately after intubation and positive end expiratory pressure (PEEP) 7 cm H20 until extubation. Inspiratory oxygen concentration 40% during recovery from anesthesia.
2. The group not receiving RM, PEEP 0 cm H2O and inspiratory oxygen concentration 100% during recovery from anesthesia.

The volume changes of the chest wall is monitored continuously by OEP, functional residual capacity (FRC) and arterial oxygenation are measured at the defined points in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ASA classification I-II, scheduled for elective surgery requiring general anesthesia
* signed informed consent

Exclusion Criteria:

* BMI > 35
* co-existing respiratory disease (COPD, asthma )
* patient refusal
* pregnancy
* deformities of the thorax

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Opto-electronic plethysmography (OEP) | 1. 5 min after each of these steps: the onset of the mechanical ventilation, the randomization, the end of the surgery 2. continuously during recovery 3. one hour after extubation
  Respiratory movements and thoracic and abdominal volume changes is recorded continuously using OEP (OEP system, BTS,Milan, Italy) by analysing the movements of retro-reflective markers using six video cameras connected to an automatic optoelectronic motion analyser.

SECONDARY OUTCOMES:
Functional residual capacity (FRC) | 5 min after each of these steps: the onset of mechanical ventilation, the randomization, the end of the sergery
Oxygenation (paO2) | 5 min after each of these steps: the onset of mechanical ventilation, the randomization, the end of the surgery, extubation
  Arterial blood gas measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Anesthesia and Intensive care dep., Uppsala, Uppsala County, Sweden